CLINICAL TRIAL: NCT03767933
Title: A Study of Non-Steroidal or Opioid Analgesia Use for Children With Musculoskeletal Injuries: The No OUCH Trials
Brief Title: Non-Steroidal or Opioid Analgesia Use for Children With Musculoskeletal Injuries
Acronym: No OUCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Manitoba (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); University of Calgary (Other); The Hospital for Sick Children (Other); University of Ottawa (Other); Western University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00073476
Record Dates: First submitted 2018-11-21; First posted 2018-12-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Musculoskeletal Injury
Keywords: Pediatrics; Emergency; Analgesia; Opioids; Combination therapy; Ibuprofen; Acetaminophen; Hydromorphone
MeSH Terms: conditions — Emergencies; Agnosia | interventions — Ibuprofen; Acetaminophen; Hydromorphone

STUDY DESIGN:
Intervention Model Description: This study will be comprised of two Phase 2, six-centre, randomized, double blind, placebo-controlled trials that will be run simultaneously. The investigators expect that the number of participants recruited and the time to completion of both trials will be more efficient as recruitment for both will occur simultaneously. They propose to conduct this study with a novel preference-informed complementary trial design, in which they will conduct two simultaneous 'sister' trials. Caregiver/child pairs presenting to the ED with acute MSK limb injury will decide in which trial they wish to participate: the Opioid trial or the Non-Opioid trial. The design of each trial will be informed by its sister, or complementary, trial. Once the caregiver/child pair has chosen their preferred trial, conduct within each trial will follow traditional randomized, double-blind placebo-controlled superiority trial methodology. Study endpoints will be identical for both trials within this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research staff, emergency department staff, and participants will be masked with respect to the allocated treatment. The data analyst will also be masked using codes that will not identify treatment groups until analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Non-Opioid Trial: Arm 1 (Active Comparator): Oral ibuprofen (10mg/kg, max 600mg) + Oral acetaminophen placebo, both administered once during the study at the time of recruitment.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen placebo
- Non-Opioid Trial: Arm 2 (Experimental): Oral ibuprofen (10mg/kg, max 600mg) + Oral acetaminophen (15mg/kg, maximum 1000mg), both administered once during the study at the time of recruitment.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- Opioid Trial: Arm 1 (Active Comparator): Oral ibuprofen (10mg/kg, max 600mg) + Oral acetaminophen placebo + Oral hydromorphone placebo, all administered once during the study at the time of recruitment.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen placebo; Drug: Hydromorphone placebo
- Opioid Trial: Arm 2 (Experimental): Oral ibuprofen (10mg/kg, max 600mg) + Oral acetaminophen (15mg/kg, maximum 1000mg) + Oral hydromorphone placebo, all administered once during the study at the time of recruitment.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Hydromorphone placebo
- Opioid Trial: Arm 3 (Experimental): Oral ibuprofen (10mg/kg, max 600mg) + Oral acetaminophen placebo + Oral hydromorphone (0.05mg/kg, maximum 5 mg), all administered once during the study at the time of recruitment.
  Interventions: Drug: Ibuprofen; Drug: Hydromorphone; Drug: Acetaminophen placebo

INTERVENTIONS:
Drug: Ibuprofen — 10mg/kg, maximum 600mg; Oral liquid
  Other Names: Advil; Motrin
Drug: Acetaminophen — 15mg/kg, maximum 1000mg; Oral liquid
  Other Names: Tylenol; Tempra
  Arms: Non-Opioid Trial: Arm 2; Opioid Trial: Arm 2
Drug: Hydromorphone — 0.05mg/kg, maximum 5 mg; Oral liquid
  Other Names: Dilaudid; pms-Hydromorphone
  Arms: Opioid Trial: Arm 3
Drug: Acetaminophen placebo — Oral liquid
  Arms: Non-Opioid Trial: Arm 1; Opioid Trial: Arm 1; Opioid Trial: Arm 3
Drug: Hydromorphone placebo — Oral liquid
  Arms: Opioid Trial: Arm 1; Opioid Trial: Arm 2

SUMMARY:
Musculoskeletal (MSK) injuries, including limb injuries, are the most common cause for Emergency Department (ED) visits for children with pain. Broken arms and legs are known to cause moderate to severe pain in most children, yet previous research shows that children's pain in the emergency department is still under-treated. Further, children are less likely to receive appropriate pain medicine than adults with similar injuries.

The purpose of this research study is to compare the effectiveness and safety of 3 different possible medication combinations, for the pain management of children with acute MSK limb injuries. The pain medicines the investigators are studying are ibuprofen (Advil/Motrin), acetaminophen (Tylenol/Tempra), and hydromorphone (Dilaudid).

This study will consist of 2 trials that will be run simultaneously. Eligible caregiver/ child pairs presenting to the emergency department with acute MSK limb injury will decide in which trial they wish to participate: the Opioid trial or the Non-Opioid trial. If they select the Non-opioid trial, they will have an equal chance of receiving either (a) Ibuprofen OR (b) Ibuprofen and acetaminophen. If they select the Opioid trial, they will have an equal chance of receiving either (a) Ibuprofen OR (b) Ibuprofen and acetaminophen OR (c) Ibuprofen and hydromorphone. Regardless of which study they choose, their child will, at minimum, receive Ibuprofen (Advil/Motrin) for their pain. All study medicines will be given in oral liquid form.

This study will help the investigators figure out which pain medicine or combination of pain medicines works best for children with limb injuries. Promotion of adequate acute pain treatment of children presenting to the ED may help prevent the known short and long-term effects of inadequately treated pain in children, including unpleasant memories, stress and anxiety upon future visits to healthcare, and compromised functional outcomes such as missed school.

DETAILED DESCRIPTION:
Rationale:

Multiple national and international organizations, including the American Academy of Pediatrics (AAP), have voiced concern over the emergency departments' (EDs) ability and willingness to provide appropriate analgesia for children's pain. Musculoskeletal (MSK) injury is a very common cause for ED visits for children with pain, with a child's risk of sustaining a fracture ranging from 27-42% by the age of 16 years. MSK injury is known to generate moderate to severe pain in most children and the ED serves as the critical entry point for these injured children. Despite three decades of pain research in this area, recent evidence confirms that ED pain management in children is still suboptimal. A retrospective cohort study of children presenting to the ED with an isolated long-bone fracture showed almost 1/3 received inadequate medication and 59% received no pain medications during the critical first hour of assessment. Previous studies have demonstrated that only 35% of children presenting to a Canadian pediatric ED with fractures or severe sprains received any analgesic. Further, a medical record review of two Canadian EDs showed unacceptably long delays in provision of initial analgesia, with children waiting a mean of 118 minutes to the provision of first analgesia.

The AAP's consensus statement on the assessment and management of pain in children recommends acetaminophen, ibuprofen, and opioids as the top three medication choices for the treatment of acute pain in children. These are also the top three most commonly used treatments in the ED for children with MSK injury pain. It stands to reason that clinicians (and certainly patients and their families) would prefer medication that has the best efficacy and safety profile. Although not based on robust evidence, there has recently been a concerted movement to limit opioid use in children. This is due, in part, to recent controversial publications and the Centre for Disease Control (CDC)'s position statement regarding opioid use in adults. Clinicians are increasingly less likely to prescribe oral opioids to younger children, and caregivers are increasingly less willing to accept or administer them.

Clinicians are currently seeking effective (and for many, non-opioid) oral analgesic options for their pediatric patients. Researchers have yet to identify the optimal acute pain management strategy for children with a suspected fracture, as very few studies of analgesic combination therapy for this injury exist, and monotherapy has been shown to be inadequate 50% of the time. This team's previous work has demonstrated that a combination of oral morphine with ibuprofen was no more effective and was less safe than oral ibuprofen, alone, for suspected fracture pain. Similarly, oxycodone was no more effective and was less safe than ibuprofen for post-discharge fracture pain. There is some emerging work from non-ED settings to suggest that oral hydromorphone may be an effective alternative to these two opioid medications. The investigators wish to study if acetaminophen or hydromorphone, when added to ibuprofen, offers more clinical pain relief than ibuprofen alone. They also wish to study if the combination of hydromorphone and ibuprofen is more clinically effective than the combination of acetaminophen with ibuprofen. This study, which will consist of two clinical trials, will inform health-care decisions by providing evidence for the effectiveness and safety of commonly prescribed analgesic combination therapies, and compare them to the most commonly used monotherapy, ibuprofen.

Methods:

This study will be comprised of two Phase 2, six-centre, randomized, double blind, placebo-controlled trials that will be run simultaneously. These two 'sister trials will be run simultaneously within this novel preference-informed complementary trial design. Caregiver/child pairs presenting to the ED with acute MSK limb injury will decide in which trial they wish to participate: the Opioid trial or the Non-Opioid trial.

Those willing to consider an Opioid will be randomized to receive either single-dose: (a) oral ibuprofen (10mg/kg, max 600mg) plus 2 placebos (both oral hydromorphone and acetaminophen), OR (b) oral ibuprofen (10mg/kg, max 600mg) + oral acetaminophen (15 mg/kg, max 1000mg) plus hydromorphone placebo OR (c) oral ibuprofen (10mg/kg) + oral hydromorphone (0.05 mg/kg, max 5 mg) plus acetaminophen placebo. Those not willing to consider an opioid will be enrolled in the Non-Opioid trial and will be randomized to receive a single dose of (a) oral ibuprofen (10mg/kg, max 600mg) + oral acetaminophen (15 mg/kg, max 1000mg) OR (b) oral ibuprofen (10mg/kg, max 600mg) + oral acetaminophen placebo. Those without a preference for either trial will be assigned to the Opioid trial, as this one includes all three options of possible medication combinations. The investigators will measure pain scores, assess safety, and acquire other study measures, at designated study time points.

ELIGIBILITY:
Inclusion Criteria:

1. Child aged 6-17 years
2. Presenting to the emergency department with an acute limb injury (<24 hours old) that is neither obviously deformed nor having neuro-vascular compromise (as assessed by the triage nurse)
3. Self-reported pain score > 5 on the 0 to 10 verbal Numerical Rating Scale at triage

Exclusion Criteria:

1. Deemed to require immediate intravenous (IV) or intranasal (IN) pain medications by the clinical team
2. Previously known hypersensitivity to study medications
3. Acetaminophen or NSAID use within 3 hours prior to recruitment
4. Opioid use within 1 hour prior to recruitment
5. Caregiver and/or child cognitive impairment precluding the ability to self-report pain or respond to study questions
6. Injury suspected to be due to non-accidental trauma/ child abuse (as assessed by the triage nurse or reported by the family)
7. Suspected multi-limb fracture
8. Chronic pain that necessitates daily analgesic use
9. Hepatic or renal disease/dysfunction
10. Bleeding disorder
11. Known pregnancy
12. Vomiting that precludes the ability to take oral medications (as determined by the family)
13. Caregiver and/or child inability to communicate fluently in English or French in the absence of a native language interpreter
14. Caregiver unavailable for follow-up
15. Previous enrolment in the NO OUCH study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 710 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
vNRS Pain Score | At 60 minutes post study drug administration (ie. T-60)
  The self-reported vNRS pain score. The 11 point 0-10 verbal Numerical Rating Scale (vNRS) is the most commonly used pain measurement tool for our study age group and has been validated in a number of children's pain studies.

SECONDARY OUTCOMES:
Pain Score <3 | At 60 minutes post study drug administration (ie. T-60)
  The proportion of patients with a vNRS pain score <3 at 60 minutes. The 11 point 0-10 verbal Numerical Rating Scale (vNRS) is the most commonly used pain measurement tool for our study age group and has been validated in a number of children's pain studies.
Pain Score Reduction of at least 2 points out of 10 | At 60 minutes post study drug administration (ie. T-60)
  The proportion of patients with a vNRS pain score reduction of at least 2 points out of 10. The 11 point 0-10 verbal Numerical Rating Scale (vNRS) is the most commonly used pain measurement tool for our study age group and has been validated in a number of children's pain studies.
Between Group Pain Scores | At 30, 60, 90, and 120 minutes post study drug administration, at Time of Medical Examination (approximately 90 minutes after time of recruitment) and at Time of X-Ray (approximately 60 minutes after time of recruitment)
  Between group differences in vNRS pain scores. The 11 point 0-10 verbal Numerical Rating Scale (vNRS) is the most commonly used pain measurement tool for our study age group and has been validated in a number of children's pain studies.
Satisfaction with Pain Relief | At the time of discharge from the emergency department (approximately 3 hours after time of recruitment)
  Self-reported caregiver and child satisfaction with pain relief and acceptability of study medications, using a previously employed 5 point Likert scale. This scale ranges from very satisfied to very dissatisfied for caregivers, and ranges from very happy to very sad for children.
Length of Stay | At the time of discharge from the emergency department (approximately 3 hours after time of recruitment)
  Emergency Department length of stay
Missed Fractures or Dislocations | In the 1 week following administration of study medication
  Frequency of missed fractures or dislocations
Additional Analgesic Requirements | In the 60 minutes following administration of study medication
  Proportion of children administered a rescue analgesic
Time to Effective Analgesia | At 30, 60, 90, and 120 minutes post study drug administration, and at the Time of Medical Examination (approximately 90 minutes after time of recruitment) and Time of X-Ray (approximately 60 minutes after time of recruitment)
  Time to effective analgesia, defined as the first vNRS pain score <3 post-intervention
VAS Pain Scores | At 30, 60, 90, and 120 minutes post study drug administration, and at the Time of Medical Examination (approximately 90 minutes after time of recruitment) and Time of X-Ray (approximately 60 minutes after time of recruitment)
  Children's self-reported pain intensity on the Visual Analog Scale (VAS). The VAS consists of a straight line with the anchor 'no pain' on one end and 'the worst imaginable pain' at the other end. It is a validated measure for the assessment of pain in children.
FPS-R Pain Scores | At 30, 60, 90, and 120 minutes post study drug administration, and at the Time of Medical Examination (approximately 90 minutes after time of recruitment) and Time of X-Ray (approximately 60 minutes after time of recruitment)
  Children's self-reported pain intensity on the Faces Pain Scale-Revised (FPS-R). The FPS-R consists of 6 faces, from left to right, each showing a greater level of pain than the previous one, with scores varying from 0 (no pain), 2, 4, 6, 8, and 10 (very much pain). The FPS-R is a validated measure for the assessment of pain in children.
Adverse Events | Up to 24 hours post study drug administration
  Proportion of children with adverse events related to study drug administration.
Serious Adverse Events | Up to 24 hours post study drug administration
  Proportion of children with any serious adverse events during the study period
RSS | At 0, 30, 60, 90, and 120 minutes post study drug administration, and at the Time of Medical Examination (approximately 90 minutes after time of recruitment) and Time of X-Ray (approximately 60 minutes after time of recruitment)
  Proportion of children in each study group with a Ramsay Sedation Score (RSS) score between 1 to 3
Specific Adverse Events | Up to 24 hours post study drug administration
  Proportion of children with each specific adverse event type during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Samina Ali, MD, Principal Investigator — University of Alberta/Stollery Children's Hospital
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital Emergency Department, Edmonton, Alberta
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - Childrens Hospital at London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the CIHR Open Access Policy. The trials will be registered at ClinicalTrials.gov, and results information from this study will be submitted to ClinicalTrials.gov. Also, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint by contacting the Women and Children's Health Research Institute (WCHRI) Data Coordinating Center (DCC). Conduct, reporting, editing, and publication of resultant scholarly work will be guided by the International Committee of Journal Medical Editors (ICJME)'s published recommendations.
  The identity of participants will not be revealed in any published data or in presentation of the information obtained as a result of this study.
Time Frame: Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint
Access Criteria: Researchers will need to contact the WCHRI DCC for access to the data

REFERENCES:
- [Derived] Ali S, Klassen TP, Candelaria P, Bhatt M, Sawyer S, Stang A, Yaskina M, Heath A, Pechlivanoglou P, Offringa M, Drendel AL, Hickes S, Poonai N; KidsCAN PERC Innovative Pediatric Clinical Trials No OUCH Study Team. Acetaminophen (Paracetamol) or Opioid Analgesia Added to Ibuprofen for Children's Musculoskeletal Injury: Two Randomized Clinical Trials. JAMA. 2026 Jan 8:e2525033. doi: 10.1001/jama.2025.25033. Online ahead of print. PMID 41505155
- [Derived] Ali S, Dworsky-Fried Z, Moir M, Bharadia M, Rajagopal M, Gouin S, Sawyer S, Pellerin S, Bourrier L, Poonai N, Stang A, Leung J, van Manen M; KidsCAN PERC Innovative Pediatric Clinical Trials No OUCH Study Team. Factors Influencing Parental Decision-Making Regarding Analgesia for Children with Musculoskeletal Injury-Related Pain: A Qualitative Study. J Pediatr. 2023 Jul;258:113405. doi: 10.1016/j.jpeds.2023.113405. Epub 2023 Apr 4. PMID 37023945
- [Derived] Heath A, Yaskina M, Hopkin G, Klassen TP, McCabe C, Offringa M, Pechlivanoglou P, Rios JD, Poonai N, Ali S; KidsCAN PERC Innovative Pediatric Clinical Trials No OUCH Study Group. Non-steroidal or opioid analgesia use for children with musculoskeletal injuries (the No OUCH study): statistical analysis plan. Trials. 2020 Sep 3;21(1):759. doi: 10.1186/s13063-020-04503-y. PMID 32883371
- [Derived] Ali S, Rajagopal M, Klassen T, Richer L, McCabe C, Willan A, Yaskina M, Heath A, Drendel AL, Offringa M, Gouin S, Stang A, Sawyer S, Bhatt M, Hickes S, Poonai N; KidsCAN PERC Innovative Pediatric Clinical Trials No OUCH Study Team. Study protocol for two complementary trials of non-steroidal or opioid analgesia use for children aged 6 to 17 years with musculoskeletal injuries (the No OUCH study). BMJ Open. 2020 Jun 21;10(6):e035177. doi: 10.1136/bmjopen-2019-035177. PMID 32565458